CLINICAL TRIAL: NCT06411847
Title: The Effectiveness of Virtual Appointments on Compliance With Twin Block Wear: A Randomised Controlled Trial
Brief Title: The Effectiveness of Virtual Appointments on Compliance With Twin Block Wear
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Dublin Dental University Hospital (Other)
Responsible Party: Principal Investigator, Abeer Hasan, Specialist Registrar in Orthodontics, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SJH/TUH JREC: 3411
Record Dates: First submitted 2024-05-03; First posted 2024-05-13 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Compliance, Patient
Keywords: Twin Block; Functional Appliances; Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Appointment Group (Experimental): This group will receive additional virtual appointments as an adjunct to standard care
  Interventions: Behavioral: Virtual appointments
- Control Group (No Intervention): The group will receive standard Care

INTERVENTIONS:
Behavioral: Virtual appointments — This group will receive the same information as the control group with additional virtual appointments at 1 week, 2 weeks and 6 weeks after fitting a Twin Block appliance. These will be scheduled and held via BlueEye Clinic (RedZinc Services Ltd.), a web-based GDPR compliant platform that allows patients to access a remote video consultation via a link sent to the participant/parent's device. The content of these appointments will follow a template that addresses the patient's experience, difficulties faced and how to overcome these, and would incorporate use of visual aids to highlight expected changes over the duration of wear. The appointments would be held in the late afternoons (after school).
  Other Names: Remote consultations
  Arms: Virtual Appointment Group

SUMMARY:
The investigators aim to determine the effect of virtual appointments on compliance with Twin Block wear. Patients satisfying the inclusion criteria requiring a Twin Block appliance will be requested to participate in the study. Those selected will be allocated to either the intervention or control group. The control group will receive routine verbal instruction and a standard information leaflet at the start of their treatment. The intervention group will additionally receive virtual appointments over the initial period of treatment involving focussed discussion on twin block wear experience and use of visual aids.

Wear time will be objectively recorded in both groups using a temperature-sensitive microsensor embedded in the Twin Block appliance, and occlusal changes will be measured at each standard recall visit. A comparison of the data obtained from each group will be undertaken to determine whether there is a significant difference in compliance with twin block wear between participants who receive adjunctive virtual appointments to those who do not.

DETAILED DESCRIPTION:
A Twin Block is a removable functional appliance commonly used in growing patients to correct a Class II malocclusion due to a combination of accelerated mandibular growth and dento-alveolar change. The Twin Block consists of two separate intersecting appliances that hold the lower jaw in a forward-postured position to correct anterior-posterior skeletal and dental relationships, thereby improving the facial profile and reducing the projection of the upper front teeth (overjet). In order to achieve these desired changes, Twin Blocks need to be worn for at least 12 hours per day. Due to the removable nature of the appliance, treatment success is reliant on patient compliance.

Compliance with twin block wear is known to be suboptimal, with non-compliance rates of up to 34% recorded in the literature. This may be attributed to several factors associated with Twin Block wear, such as lack of self-motivation, physical impairment, social concerns and forgetfulness. Virtual appointments could potentially help to address some of these issues.

Previously explored interventions to improve compliance with removable appliances include the use of calendars, known monitoring, conscious hypnosis and establishing implementation intentions. Patients have also recommended the use of visual aids, effective communication tools, positive reinforcement and reminders, all of which may be incorporated within virtual appointments, in improving compliance with Twin Block wear. The effectiveness of virtual appointments in improving Twin Block wear is yet to be assessed.

The use of remote consultation in healthcare offers potential advantages to patients, reducing travel costs and improving convenience, while also potentially enhancing cost-effectiveness and efficiency. Patients report high levels of satisfaction with virtual dental appointments related to ease of use, effectiveness and reliability. Remote communications have been employed successfully to deliver oral health advice, diagnose, monitor development, and provide behaviour guidance for paediatric patients. 'Teledentistry' has been adopted in orthodontics for remote consultations and monitoring, owing to advancements in technology, the need for social distancing during the COVID-19 pandemic, demand and convenience. Notwithstanding this, there is limited evidence available concerning its effectiveness either as a substitute to or an adjunct to conventional in-person visits.

As patients tend to over-report wear time of removable appliances, compliance is better measured objectively through the use of temperature-sensitive microsensors embedded within Twin Block appliances. These devices work by taking frequent readings of the surrounding temperature. When the temperature falls to below that of the intra-oral environment, it suggests the appliance is no longer being worn. The data collected from the sensor is interpreted through dedicated software and can be translated to the number of hours of wear per day. TheraMon® microsensors have been placed in various removable appliances to provide acceptable accuracy in measuring wear-time, with mean under-reporting of 4% and a mean difference of approximately one hour between actual and recorded wear described.

ELIGIBILITY:
Inclusion Criteria:

* Males 11-14 years old, Females 10-13 years old at start of Twin Block treatment
* Class II division 1 incisor relationship with an overjet ≥ 7mm
* Access to a smartphone with a microphone and camera
* Willingness to participate in the study

Exclusion Criteria:

- Patients receiving treatment with fixed appliances in conjunction with Twin Block treatment

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Wear Time | Data will be collected at standard in-person recall visits at 1 month, 3 month and 6 months.
  Wear time in minutes will be recorded by a Theramon® microsensor (Handelsagentur Gschladt, Hargelsberg, Austria, or Forestadent, Pforzheim, Germany) embedded in the maxillary appliance, supplemented with a self-completed wear chart.

SECONDARY OUTCOMES:
Occlusal change | Data will be collected at standard in-person recall visits at 1 month, 3 month and 6 months.
  Measurement of overjet in millimetres

CONTACTS AND LOCATIONS:
Locations (2):
- Ireland (2):
  - HSE Orthodontic Unit, Loughlinstown, Dublin
  - HSE Orthodontic Unit, Tallaght, Dublin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brierley CA, Benson PE, Sandler J. How accurate are TheraMon(R) microsensors at measuring intraoral wear-time? Recorded vs. actual wear times in five volunteers. J Orthod. 2017 Dec;44(4):241-248. doi: 10.1080/14653125.2017.1365220. Epub 2017 Aug 22. PMID 28826346
- [Background] Al-Moghrabi D, Salazar FC, Pandis N, Fleming PS. Compliance with removable orthodontic appliances and adjuncts: A systematic review and meta-analysis. Am J Orthod Dentofacial Orthop. 2017 Jul;152(1):17-32. doi: 10.1016/j.ajodo.2017.03.019. PMID 28651764
- [Background] Park JH, Kim JH, Rogowski L, Al Shami S, Howell SEI. Implementation of teledentistry for orthodontic practices. J World Fed Orthod. 2021 Mar;10(1):9-13. doi: 10.1016/j.ejwf.2021.01.002. Epub 2021 Feb 25. PMID 33642260